CLINICAL TRIAL: NCT02562183
Title: The Study to Reevaluate the Safety and Efficacy of Human Urinary Kallikrein
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Techpool Bio-Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KLK-4002
Record Dates: First submitted 2015-09-10; First posted 2015-09-29 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Cerebral Infarction
MeSH Terms: conditions — Cerebral Infarction | interventions — Kallikreins; Tissue Kallikreins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- kallikrein group (Experimental): Subjects receive kallikrein treatment according to real clinical practice (suggest above 14days treatment),0.15 peptide nucleic acids(PNA), once a day.
  Interventions: Drug: kallikrein

INTERVENTIONS:
Drug: kallikrein — Using kallikrein
  Other Names: KLK; Human urinary kallikrein

SUMMARY:
In order to reevaluate safety and efficacy of human urinary kallikrein in treating acute cerebral infarction ,a multi-center, open label , single group study was designed. Expect to enroll 60 sites and 2186 subjects. Subjects will receive kallikrein treatment according to real clinical practice (suggest above 14days treatment) and 90 days follow up

ELIGIBILITY:
Inclusion Criteria:

1. Acute anterior circulation cerebral infarction diagnosed ≤ 48h;
2. First time diagnosed or have history of acute anterior circulation cerebral infarction without serious sequelae(mRS=0-2);
3. Age from 18 to 80 years old;
4. National Institute of Health stroke scale(NIHSS) from 6 to 25;
5. Have provided signed written informed consent from the patient or the patient's legal representative.

Exclusion Criteria:

1. Brain CT shows cerebral hemorrhage disease: cerebral hemorrhage, subarachnoid hemorrhage, etc.
2. Transient ischemic attack(TIA);
3. Serious disturbance of consciousness: Glasgow Coma ScaleGCS（GCS）≤8;
4. Combined angiotensin-converting enzyme inhibitor(ACEI) less than 5 half-time(according to its instruction), or need to be treated with ACEI;
5. Cases treated with thrombolysis / stent surgery or expected to be treated with thrombolysis / interventional therapy / stent surgery.
6. subjects with bleeding disorders at Past or present, laboratory tests: INR > 1.5 or APTT > 2 times;
7. subjects with abnormal liver function (ALT/AST > 1.5 * ULN) and abnormal renal function (Cr> normal upper limit);
8. subjects with history of epilepsy or other serious systemic disease before onset of AIS refused by PI to enroll ;
9. subjects with cardiogenic stroke or cardiogenic stroke related high-risk factors identified by PI, such as atrial fibrillation, echocardiography or Mural thrombus etc;
10. subjects diagnosised any malignancy (except basal cell carcinoma) within 5 years prior to the start of the study;
11. subjects with severe dementia or can't cooperate to evaluate identified by PI;
12. suffering from severe hypertension and failed to control :systolic blood pressure ≥200mmHg (26.6kPa) or diastolic blood pressure ≥110mmHg (14.6kPa); hypotension: systolic blood pressure< 90mmHg and/or diastolic blood pressure< 60mmHg
13. subjects be allergic or intolerant to kallikrein at past;
14. subjects be pregnant/lactating or possibly and planned pregnant;
15. subjects be unsuitable for this clinical study identified by PI.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2186 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-11-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | From enrolled to the day 90

SECONDARY OUTCOMES:
Cerebral infarction on the National Institute of Health stroke scale | The day 8,15 and 22 after enrolled
Recurrence rate of acute cerebral infarction | From enrolled to the day 90
Activities of daily living on the Barthel Index | The day 15,22 and 90 after enrolled
Patients body status on the Modified Rankin Scale | The day 15, 22 and 90 after enrolled
EQ-5D-3L score | The day 15, 22 and 90 after enrolled
Evaluation of pharmaceutical economics | The day 15, 22 and 90 after enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Liying Cui, Doctor, Principal Investigator — Peking Union Medical College Hospital
Locations (7):
- China (7):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - NO.2 Hospital XiaMen, Xiamen, Fujian
  - HanDan Central Hospital, Handan, Hebei
  - Harrison International Peace Hospital, Hengshui, Hebei
  - Chenzhou NO.1 People's Hospital, Chenzhou, Hunan
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The Fourth Affiliated hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ni J, Qu J, Yao M, Zhang Z, Zhong X, Cui L; RESK investigators. Re-evaluate the Efficacy and Safety of Human Urinary Kallidinogenase (RESK): Protocol for an Open-Label, Single-Arm, Multicenter Phase IV Trial for the Treatment of Acute Ischemic Stroke in Chinese Patients. Transl Stroke Res. 2017 Aug;8(4):341-346. doi: 10.1007/s12975-017-0527-5. Epub 2017 Mar 6. PMID 28265861